CLINICAL TRIAL: NCT07355608
Title: Prediction of Difficult Videolaryngoscopic Intubation and Development of a Dedicated Glottic View Score: A Multicentre Prospective Study
Brief Title: Videolaryngoscopic Difficult ıntubation and Glottic View Score: A Multicentre Prospective Study
Acronym: VIDIGLOV
Status: Not yet recruiting | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Professor of Anesthesiology, Diskapi Teaching and Research Hospital
Other Study IDs: Etlik City Hospital
Record Dates: First submitted 2025-12-02; First posted 2026-01-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Airway Management
Keywords: Airway management; Videolaryngoscope; Difficult airway

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Videolaryngoscopy has improved glottic visualization and facilitated tracheal intubation. However, difficulties-including failed intubation-still occur. At present, no prospectively derived classification system exists to assess the difficulty of videolaryngoscopic (VL) intubation across both normal and anticipated difficult airways. Additionally, current glottic view grading systems, designed for direct laryngoscopy, may not adequately capture the specific challenges of VL intubation.

Objectives:

This study aims to:

1. Develop a predictive model for difficult VL intubation in surgical patients with both normal and anticipated difficult airways.
2. Create a glottic view scoring system specifically tailored to videolaryngoscopy.
3. Compare the predictive accuracy of the new scoring system with existing laryngeal view grades in forecasting difficult VL intubation.

DETAILED DESCRIPTION:
Background:

Videolaryngoscopy has improved glottic visualization and facilitated tracheal intubation. However, difficulties-including failed intubation-still occur. At present, no prospectively derived classification system exists to assess the difficulty of videolaryngoscopic (VL) intubation across both normal and anticipated difficult airways. Additionally, current glottic view grading systems, designed for direct laryngoscopy, may not adequately capture the specific challenges of VL intubation.

Objectives:

This study aims to:

1. Develop a predictive model for difficult VL intubation in surgical patients with both normal and anticipated difficult airways.
2. Create a glottic view scoring system specifically tailored to videolaryngoscopy.
3. Compare the predictive accuracy of the new scoring system with existing laryngeal view grades in forecasting difficult VL intubation.

Methods:

A prospective cohort of 4,977 patients will be enrolled. Patient and intubation related variables-including VL findings, airway features, clinical parameters, device, and procedural details-will be analyzed. Binary logistic regression will be employed to build the initial predictive model. In parallel, machine learning techniques (Random Forest, Support Vector Machine, XGBoost, LightGBM, etc.) will be applied to evaluate predictive performance. Comparative analysis will be conducted between the machine learning models and the logistic regression baseline.

Expected Impact:

The development of a robust predictive tool and an associated VL-specific glottic view score could enhance clinical decision making, particularly in identifying patients at risk of difficult or failed VL intubation. This may support early consideration of awake tracheal intubation, and use of standardized terminology and reduce complications associated with difficult airway management

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Both with normal or predicted difficult airways
* Undergoing orotracheal intubation with a videolarygoscope

Exclusion Criteria:

* Rapid sequence intubation
* Double lumen tube intubation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, both with normal or predicted difficult airways, undergoing orotracheal intubation with a videolarygoscope, for a case mix of surgeries
Sampling Method: Probability Sample
Enrollment: 4977 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Failed first intubation attempt | 2 minutes after anesthesia induction
  Failed to intubate at firtst attempt
Difficult intubation | 2 minutes after anesthesia induction
  Failed to intubate at 1-2 attempts and/or intubation duration longer than 120 second
Failed intubation | 2 minutes after anesthesia induction
  Not able to intubate the patient
Intubation duration | 2 minutes after anesthesia induction
  Time elapsed from entring the blade between the teeth to detecting an entidal carbondioxide trace
Glottic view description | 2 minutes after anesthesia induction
  Vocal cords are fully visible Vocal cords are partially separately Vocal cords are not visible Cords are adducted Epiglottis is visible Epiglottis is large Epiglottis is small Epiglottis is edematous Epiglottis mass is present Arytenoids are visible Arytenoid luxation or subluxation Arytenoid edema Valecula problem (edema, Coffee grounds, etc., unable to insert a blade) Aryepiglottic plica pathology (edema, Coffee grounds scar) Laryngeal structures should be formed Glottic stenosis Laryngospasm

SECONDARY OUTCOMES:
Percentil of glottic opening score | 2 minutes after anesthesia induction
  the percentage of glottic opening seen, defined by the linear span from the anterior commissure to the inter-arytenoid notch
Cormack lehanne score | 2 minutes after anesthesia induction
  grade 1 being a full view of the glottis, grade 2 being a partial view, grade 3 being only a view of the epiglottis, and grade 4 being an absent view of the glottis and epiglottis

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Yazıcıoğlu Ünal, professor, Principal Investigator — Ankara Etlik City Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Etlik City Hospital, Ankara
  - Akdeniz University Medical Faculty, Antalya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xia M, Jin C, Zheng Y, Wang J, Zhao M, Cao S, Xu T, Pei B, Irwin MG, Lin Z, Jiang H. Deep learning-based facial analysis for predicting difficult videolaryngoscopy: a feasibility study. Anaesthesia. 2024 Apr;79(4):399-409. doi: 10.1111/anae.16194. Epub 2023 Dec 13. PMID 38093485
- [Background] O'Loughlin EJ, Swann AD, English JD, Ramadas R. Accuracy, intra- and inter-rater reliability of three scoring systems for the glottic view at videolaryngoscopy. Anaesthesia. 2017 Jul;72(7):835-839. doi: 10.1111/anae.13837. Epub 2017 Mar 24. PMID 28337769